CLINICAL TRIAL: NCT04101422
Title: Utilizing Augmented Reality as an Adjunct for Smoking Cessation; Development and Initial Validation
Brief Title: Utilizing Augmented Reality as an Adjunct for Smoking Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MCC-20007; R34DA047598-03 (NIH)
Record Dates: First submitted 2019-09-23; First posted 2019-09-24 (Actual); Results first posted 2023-05-22 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-04

CONDITIONS: Smoking
Keywords: Quit Smoking; Augmented Reality; Smoking
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Development of Augmented Reality (AR) Application (No Intervention): Investigators will collaborate with an AR software specialist to develop AR stimuli that are embedded within a basic digital application.
- Pilot Testing of AR Application (Experimental): AR stimuli (smoking, e.g, cigarette, ashtray, lighter; and non-smoking, e.g., pen, notebook, eraser) will be piloted on a small group of smokers to receive feedback and modify as needed. Participants will answer questions from a 10 point Likert scale that will asses urge from 1 (absolutely no urge to smoke) to 10 (strongest urge to smoke) and reality/co-existence (how realistic the item looks, and it's integration into the environment), from 1 (Not at all) to 10 (Very Much). Participants will then be asked additional open-ended questions about the quality of the images following the ratings of the images.
  Interventions: Behavioral: Augmented Reality 1
- Laboratory Validation of AR Stimuli Session 1: Cue Reactivity (Experimental): Participants will attend 1st lab based session that will test cue-reactivity. Participant will be randomized to view either AR images, or in vivo items first. Order of presentation of items will also be randomized within the type (AR or in vivo).Session 1 should last under 1 hour.
  Interventions: Behavioral: Augmented Reality 2
- Laboratory Validation of AR Stimuli Session 2: Extinction (Experimental): Participants will be randomized into either the extinction or control group. 28 trials of AR cues will be presented for each group. Both groups will receive the same neutral cue in Trial 1 (to establish baseline urge) and the same smoking cue in Trial 2 (for pre-test cue-reactivity). The extinction group will receive smoking cues for trials 3-26, whereas the control group will receive neutral cues. Both groups will receive matched smoking cues for trial (27) followed by matched neutral cues for the final trial (28), for post-test cuereactivity. Each cue will be presented for 1 minute and will be shown 4 times in trials 3-26. Following each cue, participants will complete the single-item measure of urge. Following the final trial (28) for both groups, participants will be presented with one of their own cigarettes and asked to take at least one puff. Latency to smoke will later be determined using time stamps on the video recording. Session 2 is expected to last 1.25 hours.
  Interventions: Behavioral: Augmented Reality 4
- Testing AR Application (Experimental): Participants will be instructed to use the AR app that presents smoking-related stimuli (cigarette, ashtray, lighter) in locations/situations where they typically smoke with the goal of at least 5 uses per day for 7 days. Usage and rating data will be collected in real-time. Participants will also be asked to rate their urge to smoke on the smartphone app at selected times. Participants will complete a telephone interview to provide additional feedback on the app, answer questions related to smoking behavior, and receive an in-person interview on their perceptions of the app as a potential cessation tool. Participants will use the smart phone application for 7 days.
  Interventions: Behavioral: Augmented Reality 3

INTERVENTIONS:
Behavioral: Augmented Reality 1 — Participants will use an Augmented Reality (AR) application on smart phones. The AR application will create simulated examples of AR stimuli (cigarettes, lighters, ashtrays) and non-smoking related stimuli (pens, notebook, eraser).
  Arms: Pilot Testing of AR Application
Behavioral: Augmented Reality 2 — Participants will use an Augmented Reality (AR) application on smart phones. The AR application will create simulated examples of smoking related AR stimuli (cigarettes, lighters, ashtrays) as well as non-smoking images (pens, notebook, etc.). They will also be presented with real smoking (e.g., ashtray) and non-smoking (e.g., pencil) items. Their urge to smoke rating following each presentation will be compared for AR images vs. vivo items, and smoking-related vs. non-smoking related.
  Arms: Laboratory Validation of AR Stimuli Session 1: Cue Reactivity
Behavioral: Augmented Reality 3 — Participants will use an Augmented Reality )AR) application on smart phones in locations and situations where they typically smoke. the application will create simulated examples of AR stimuli (cigarettes, lighters, ashtrays). Participants will have a goal of using application at least 5 times per day for 7 days. Usage and rating data will be collected in real-time.
  Arms: Testing AR Application
Behavioral: Augmented Reality 4 — Participants will use an Augmented Reality (AR) application on smart phones. The AR application will create simulated examples of AR stimuli (cigarettes, lighters, ashtrays) as well as non-smoking images (pens, notebook, etc.) Their urge to smoke rating following each presentation will be compared from baseline urge to smoke. The post-test urge to smoke will be compared between control group and extinction group.
  Arms: Laboratory Validation of AR Stimuli Session 2: Extinction

SUMMARY:
The purpose of the study is to develop an preliminary test a tobacco smoking-related augmented reality (AR) paradigm for eventual development as an adjunctive tobacco cessation intervention.

ELIGIBILITY:
Inclusion Criteria:

* Currently smoking ≥ 3 cigarettes per day for the past year
* Breath carbon monoxide (CO) level ≥ 5 ppm
* Motivated to quit smoking
* Aim 1 & 2 Only: Valid home address in the Tampa Bay area
* Functioning telephone number
* Can speak, read, and write in English
* Aim 3: Must have a smartphone that participant is willing to use during the study
* Aim 3: Motivated to quit smoking within the next month

Exclusion Criteria:

* Regular use (e.g., no more than 1/3 of month) of other tobacco products (cigars)
* Household member already enrolled in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2019-10-07 (Actual); Primary Completion 2022-02-14 (Actual); Study Completion 2022-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Vinci, Ph.D., Principal Investigator — Moffitt Cancer Center; Thomas Brandon, Ph.D., Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Brandon KO, Vinci C, Kleinjan M, Hernandez LM, Sawyer LE, Sutton SK, Brandon TH. Testing Augmented Reality for Eliciting Cue-Provoked Urges to Smoke: Toward Moving Cue-Exposure Into the Real World. Nicotine Tob Res. 2021 May 4;23(5):861-865. doi: 10.1093/ntr/ntaa259. PMID 33277653
- [Derived] Yang MJ, Brandon KO, Sutton SK, Kleinjan M, Sawyer LE, Brandon TH, Vinci C. Augmented reality as a novel approach for addiction treatment: development of a smoking cessation app. Ann Med. 2022 Dec;54(1):3096-3106. doi: 10.1080/07853890.2022.2140451. PMID 36345961
- [Derived] Yang MJ, Brandon KO, Sutton SK, Kleinjan M, Hernandez LM, Sawyer LE, Brandon TH, Vinci C. Augmented reality for extinction of cue-provoked urges to smoke: Proof of concept. Psychol Addict Behav. 2022 Dec;36(8):990-998. doi: 10.1037/adb0000868. Epub 2022 Jul 14. PMID 35834198

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The 17 participants in the Laboratory Validation of AR Stimuli Session 1: Cue Reactivity group were then randomized into either the Laboratory Validation of AR Stimuli Session 2: Extinction group or Control group.
Groups:
- Laboratory Validation of AR Stimuli Session 2: Extinction or Control: Participants will be randomized into either the extinction or control group. 28 trials of AR cues will be presented for each group. Both groups will receive the same neutral cue in Trial 1 (to establish baseline urge) and the same smoking cue in Trial 2 (for pre-test cue-reactivity). The extinction group will receive smoking cues for trials 3-26, whereas the control group will receive neutral cues. Both groups will receive matched smoking cues for trial (27) followed by matched neutral cues for the final trial (28), for post-test cuereactivity. Each cue will be presented for 1 minute and will be shown 4 times in trials 3-26. Following each cue, participants will complete the single-item measure of urge. Following the final trial (28) for both groups, participants will be presented with one of their own cigarettes and asked to take at least one puff. Latency to smoke will later be determined using time stamps on the video recording. Session 2 is expected to last 1.25 hours.
  Augmented Reality 4: Participants will use an Augmented Reality (AR) application on smart phones. The AR application will create simulated examples of AR stimuli (cigarettes, lighters, ashtrays) as well as non-smoking images (pens, notebook, etc.) Their urge to smoke rating following each presentation will be compared from baseline urge to smoke. The post-test urge to smoke will be compared between control group and extinction group.
Period: Overall Study
Arm/Group | Pilot Testing of AR Application | Laboratory Validation of AR Stimuli Session 1: Cue Reactivity | Laboratory Validation of AR Stimuli Session 2: Extinction or Control | Testing AR Application
Started | 11 | 17 | 126 | 43
Extinction Group | 0 | 10 (10 participants were randomized to Session 2: Extincion group after completing Session 1: Cue Reactivity) | 59 (59 participants were randomized and started in the Extinction group and 5 did not complete) | 0
Control Group | 0 | 7 (7 participants were randomized to Session 2: Control group after completing Session 1: Cue Reactivity) | 67 (67 participants were randomized to the Control group and 9 did not complete.) | 0
Completed | 10 | 17 | 112 | 23
Not Completed | 1 | 0 | 14 | 20
Not completed — Ineligible | 1 | 0 | 9 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0
Not completed — Not attending to the stimuli | 0 | 0 | 4 | 0
Not completed — Did not download app | 0 | 0 | 0 | 17
Not completed — Did not use app on 4 or more occasions per protocol | 0 | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Population: Baseline Measures were not collected per intervention for Laboratory Validation of AR Stimuli Session 2: Extinction or Control. Participants in the Laboratory Validation of AR Stimuli Session 1: Cue Reactivity group were randomized into the Laboratory Validation of AR Stimuli Session 2: Extinction or Control group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pilot Testing of AR Application | Laboratory Validation of AR Stimuli Session 1: Cue Reactivity | Laboratory Validation of AR Stimuli Session 2: Extinction or Control | Testing AR Application | Total
Number analyzed (Participants) | 11 | 17 | 126 | 43 | 197
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 17 | 117 | 42 | 187
  >=65 years | 0 | 0 | 9 | 1 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 12 | 61 | 27 | 104
  Male | 7 | 5 | 65 | 16 | 93
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 8 | 5 | 16
  Not Hispanic or Latino | 9 | 16 | 117 | 38 | 180
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 2 | 2 | 4
  Black or African American | 4 | 8 | 45 | 10 | 67
  White | 7 | 9 | 78 | 29 | 123
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 11 | 17 | 126 | 43 | 197

OUTCOME MEASURES:

1. Primary Outcome: Urge to Smoke - Pilot Testing
Description: Participants will rate their urge to smoke on a 10-point Likert scale from 1 (absolutely no urge to smoke) to 10 (strongest urge to smoke).
Time Frame: Post-cue presentation on Day 1, immediately following cue presentation
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Pilot Testing of AR Application
Number analyzed (Participants) | 10
score on a scale
  Smoking Stimuli | 4.58 [1 to 10]
  Neutral Stimuli | 1.42 [1 to 10]

2. Primary Outcome: Urge to Smoke - AR Stimuli Session 1
Description: as for outcome 1
Time Frame: Post-cue presentation on Day 1, immediately following cue presentation
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Laboratory Validation of AR Stimuli Session 1: Cue Reactivity
Number analyzed (Participants) | 17
score on a scale
  Smoking Related AR Images | 7.50 [1 to 10]
  Neutral Images | 3.33 [1 to 10]

3. Primary Outcome: Urge to Smoke - AR Stimuli Session 2
Description: as for outcome 1
Time Frame: Post-cue presentation on Day 1, immediately following cue presentation
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Laboratory Validation of AR Stimuli Session 2: Extinction
Number analyzed (Participants) | 129
score on a scale
  Extinction condition | 5.3 (2.9)
  Control condition | 6.4 (3.3)

4. Primary Outcome: Urge to Smoke - Testing AR Application
Description: as for outcome 1
Time Frame: Day 1 - First Day of App Use, immediately following cue presentation
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Testing AR Application
Number analyzed (Participants) | 23
score on a scale | 7.61 [1 to 10]

5. Primary Outcome: Urge to Smoke - Testing AR Application
Description: as for outcome 1
Time Frame: Up to Day 7 - Last Day of App Use, immediately following cue presentation
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Testing AR Application
Number analyzed (Participants) | 23
score on a scale | 7.28 [1 to 10]

6. Secondary Outcome: Reality/Co-Existence - Pilot Testing
Description: Three items will be used to assess the quality of the AR experience. Reality (How real did the object seem to you?) Environment Co-Existence (How well did the the object appear to be part of the scene?) and User Co-Existence (How much did you feel the object was right there in front of you?). These 3 items will be assessed using a 10 point Likert Scale from from 1 (Not at all) to 10 (Very much).
Time Frame: Day 1, immediately following cue presentation
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pilot Testing of AR Application
Number analyzed (Participants) | 10
score on a scale
  Realistic | 6.49 (3.11)
  Environmental Coexistence | 6.93 (3.04)
  User Coexistence | 6.38 (3.27)

7. Secondary Outcome: Reality/Co-Existence - AR Stimuli Session 1
Description: as for outcome 6
Time Frame: Day 1, immediately following cue presentation
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Laboratory Validation of AR Stimuli Session 1: Cue Reactivity
Number analyzed (Participants) | 17
score on a scale
  Realism | 7.83 [1 to 10]
  Environmental Coexistence | 7.83 [1 to 10]
  User Coexistence | 7.17 [1 to 10]

8. Secondary Outcome: Reality/Co-Existence - AR Stimuli Session 2
Description: as for outcome 6
Time Frame: Day 1, immediately following cue presentation
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Laboratory Validation of AR Stimuli Session 2: Extinction
Number analyzed (Participants) | 129
score on a scale
  Realism | 7.91 (1.88)
  Enviromental Coexistence | 7.96 (2.31)
  User Coexistence | 8.04 (2.12)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the first day of being on study until participant was off study, an average of 5 days
Description: No Adverse Events
Arm/Group | Pilot Testing of AR Application | Laboratory Validation of AR Stimuli Session 1: Cue Reactivity | Laboratory Validation of AR Stimuli Session 2: Extinction | Testing AR Application
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/17 | 0/126 | 0/43
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/17 | 0/126 | 0/43
Other Adverse Events (participants affected / at risk) | 0/11 | 0/17 | 0/126 | 0/43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-11-23): https://cdn.clinicaltrials.gov/large-docs/22/NCT04101422/Prot_SAP_000.pdf
  • Informed Consent Form (2021-06-23): https://cdn.clinicaltrials.gov/large-docs/22/NCT04101422/ICF_001.pdf